CLINICAL TRIAL: NCT05295407
Title: Observational and Prospective Study on the Performance of Inherited Risk Assessment for Predicting Prostate Cancer From Prostate Biopsy (GenBx)
Brief Title: Performance of Inherited Risk Assessment for Predicting Prostate Cancer From Prostate Biopsy
Acronym: GenBx
Status: Recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: Northwestern University (Other); Johns Hopkins University (Other); GoPath Diagnostics (Unknown)
Responsible Party: Principal Investigator, Jianfeng Xu, Director of Program for Personalized Cancer Care, Endeavor Health
Other Study IDs: EH21-338; EH21-338 (Other: NorthShoreUH)
Record Dates: First submitted 2021-12-13; First posted 2022-03-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate biopsy; prostate cancer; inherited risk assessment; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men 40-69 years old: Men with moderately-elevated PSA (2.5-10 ng/mL) undergoing prostate biopsy for detecting prostate cancer at NorthShore University HealthSystem, Northwestern University, or Johns Hopkins Hospital. The trial will not alter any clinical practice for diagnostic biopsy that includes state-of-the-art procedures (transperineal fusion biopsy, multiparametric MRI, and novel biomarkers).
  Interventions: Genetic: Genetic Assessment

INTERVENTIONS:
Genetic: Genetic Assessment — The trial is to observe whether inherited risk, including rare pathogenic mutations (RPMs) in several major genes and SNPs-based genetic risk scores (GRS), is correlated with prostate cancer detection rate from diagnostic prostate biopsy.

SUMMARY:
Condition: Prostate cancer Intervention: Biopsy and inherited risk assessment

DETAILED DESCRIPTION:
Inherited genetic changes, including rare pathogenic mutations (RPMs) in several major genes and single nucleotide polymorphisms (SNPs)-based genetic risk scores (GRS) have been consistently associated with prostate cancer (PCa) risk. Furthermore, results from retrospective analyses of two clinical trials (PCPT and REDUCE) and biopsy cohorts revealed Caucasian men with higher GRS are 1) more likely to have positive biopsy and 2) have higher number of positive biopsy cores. These findings suggest inherited risk assessment may have clinical utility in identifying men who have a higher likelihood of positive results from diagnostic prostate biopsy. The objective of this observational trial is to confirm the clinical utility of both RPMs and GRS in a prospective study of multi-racial patients. Results from this trial will provide a critical piece of evidence for guideline committees to consider the adoption of inherited risk assessment in decision making for prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing prostate biopsy for detection of prostate cancer
* Aged 40 to 69 years
* Four ethnicity groups (Caucasian, African Americans, East Asians, Latinos)
* PSA between 2.5-10 ng/mL

Exclusion Criteria:

* Previous diagnosis of prostate cancer.
* Ethnicity outside the inclusion criterion (including mixed ethnicity).
* Any prior PSA test result outside the range of inclusion criterion.

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with moderately-elevated PSA (2.5-10 ng/mL) undergoing prostate biopsy for detecting prostate cancer at NorthShore University HealthSystem, Johns Hopkins Hospital, and Northwestern University.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer Diagnosis from Prostate Biopsy Report | 4 years
  The primary outcome measure is prostate cancer diagnosis from the prostate biopsy report. The primary goal is to compare prostate cancer detection rate in patients of three inherited risk groups (high-risk, intermediate-risk, and low-risk).

SECONDARY OUTCOMES:
The first type of secondary outcome measures is demographic key clinical variables from chart review, including | 4 years
  * Age of the patient at recruitment, measured in years
  * Ethnicity, which will be reported as either Hispanic or Latino, or not Hispanic or Latino
  * Race, which will be reported as Black/African American, East Asian, White, or Other
  * Most recent body mass index (BMI), which height and weight will be combined and reported in kg/m^2
  * Most recent PSA test result prior to prostate biopsy, which will be reported in ng/mL
  * Most recent prostate health index (PHI), which is a combination of three PSA-based blood tests that estimates the probability of having detectable prostate cancer
  * TRUS prostate volume, based on the height, length, and width of the prostate and will be reported in mL
The second type of secondary outcome measures is results from multi-parametric Magnetic Resonance Imaging (mpMRI), including | 4 years
  * Prostate total volume, measured in mL
  * Overall Prostate Imaging Reporting and Data System (PI-RAD) score, which assesses risk of clinically significant cancer being present or absent
  * Extraprostatic extension, which will be reported as present or absent
  * Seminal vesicle invasion, which will be reported as present or absent
  * Lymph node enlargement, which will be reported as present or absent
  * MRI bone metastasis, which will be reported as present or absent
  * Number of lesions, which will be reported as a numerical value
  * For each lesion, location of lesion, which will be reported as the anatomical region of the prostate where the lesion is present
  * For each lesion, size of lesion, measured in mm
  * For each lesion, PIRAD score of lesion, which assesses risk of clinically significant cancer being present or absent in the lesion
The third type of secondary outcome measures is pathological variables from prostate biopsy, including | 4 years
  * Type of prostate biopsy that was performed on the patient, which will be reported as either transperineal (TP) or transrectal ultrasound (TRUS)
  * Number of cores positive, which will be reported as a numerical value
  * Number of cores examined, which will be reported as a numerical value
  * Overall Gleason score (primary), which predicts cancer aggressiveness and prognosis
  * Overall Gleason score (secondary), which predicts cancer aggressiveness and prognosis
  * For each core, length of core, measured in cm
  * For each core, length of tumor, measured in mm
  * For each core, % of core positive, which will be reported as a numerical value as a percentage
  * For each core, % Gleason 4
  * For each core, presence of perineural invasion (PNI), will be reported as Yes or No
  * For each core, presence of cribriform, will be reported as Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Xu, MD, Dr.PH, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to release de-identified genomic and clinical data for approved researchers to replicate study or use for other discoveries.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after the study (after analysis) indefinitely
Access Criteria: With approval, researchers will be able to access published, de-identified data.

REFERENCES:
- [Background] Pritchard CC, Mateo J, Walsh MF, De Sarkar N, Abida W, Beltran H, Garofalo A, Gulati R, Carreira S, Eeles R, Elemento O, Rubin MA, Robinson D, Lonigro R, Hussain M, Chinnaiyan A, Vinson J, Filipenko J, Garraway L, Taplin ME, AlDubayan S, Han GC, Beightol M, Morrissey C, Nghiem B, Cheng HH, Montgomery B, Walsh T, Casadei S, Berger M, Zhang L, Zehir A, Vijai J, Scher HI, Sawyers C, Schultz N, Kantoff PW, Solit D, Robson M, Van Allen EM, Offit K, de Bono J, Nelson PS. Inherited DNA-Repair Gene Mutations in Men with Metastatic Prostate Cancer. N Engl J Med. 2016 Aug 4;375(5):443-53. doi: 10.1056/NEJMoa1603144. Epub 2016 Jul 6. PMID 27433846
- [Background] Na R, Zheng SL, Han M, Yu H, Jiang D, Shah S, Ewing CM, Zhang L, Novakovic K, Petkewicz J, Gulukota K, Helseth DL Jr, Quinn M, Humphries E, Wiley KE, Isaacs SD, Wu Y, Liu X, Zhang N, Wang CH, Khandekar J, Hulick PJ, Shevrin DH, Cooney KA, Shen Z, Partin AW, Carter HB, Carducci MA, Eisenberger MA, Denmeade SR, McGuire M, Walsh PC, Helfand BT, Brendler CB, Ding Q, Xu J, Isaacs WB. Germline Mutations in ATM and BRCA1/2 Distinguish Risk for Lethal and Indolent Prostate Cancer and are Associated with Early Age at Death. Eur Urol. 2017 May;71(5):740-747. doi: 10.1016/j.eururo.2016.11.033. Epub 2016 Dec 15. PMID 27989354
- [Background] Carter HB, Helfand B, Mamawala M, Wu Y, Landis P, Yu H, Wiley K, Na R, Shi Z, Petkewicz J, Shah S, Fantus RJ, Novakovic K, Brendler CB, Zheng SL, Isaacs WB, Xu J. Germline Mutations in ATM and BRCA1/2 Are Associated with Grade Reclassification in Men on Active Surveillance for Prostate Cancer. Eur Urol. 2019 May;75(5):743-749. doi: 10.1016/j.eururo.2018.09.021. Epub 2018 Oct 8. PMID 30309687
- [Background] Schumacher FR, Al Olama AA, Berndt SI, Benlloch S, Ahmed M, Saunders EJ, Dadaev T, Leongamornlert D, Anokian E, Cieza-Borrella C, Goh C, Brook MN, Sheng X, Fachal L, Dennis J, Tyrer J, Muir K, Lophatananon A, Stevens VL, Gapstur SM, Carter BD, Tangen CM, Goodman PJ, Thompson IM Jr, Batra J, Chambers S, Moya L, Clements J, Horvath L, Tilley W, Risbridger GP, Gronberg H, Aly M, Nordstrom T, Pharoah P, Pashayan N, Schleutker J, Tammela TLJ, Sipeky C, Auvinen A, Albanes D, Weinstein S, Wolk A, Hakansson N, West CML, Dunning AM, Burnet N, Mucci LA, Giovannucci E, Andriole GL, Cussenot O, Cancel-Tassin G, Koutros S, Beane Freeman LE, Sorensen KD, Orntoft TF, Borre M, Maehle L, Grindedal EM, Neal DE, Donovan JL, Hamdy FC, Martin RM, Travis RC, Key TJ, Hamilton RJ, Fleshner NE, Finelli A, Ingles SA, Stern MC, Rosenstein BS, Kerns SL, Ostrer H, Lu YJ, Zhang HW, Feng N, Mao X, Guo X, Wang G, Sun Z, Giles GG, Southey MC, MacInnis RJ, FitzGerald LM, Kibel AS, Drake BF, Vega A, Gomez-Caamano A, Szulkin R, Eklund M, Kogevinas M, Llorca J, Castano-Vinyals G, Penney KL, Stampfer M, Park JY, Sellers TA, Lin HY, Stanford JL, Cybulski C, Wokolorczyk D, Lubinski J, Ostrander EA, Geybels MS, Nordestgaard BG, Nielsen SF, Weischer M, Bisbjerg R, Roder MA, Iversen P, Brenner H, Cuk K, Holleczek B, Maier C, Luedeke M, Schnoeller T, Kim J, Logothetis CJ, John EM, Teixeira MR, Paulo P, Cardoso M, Neuhausen SL, Steele L, Ding YC, De Ruyck K, De Meerleer G, Ost P, Razack A, Lim J, Teo SH, Lin DW, Newcomb LF, Lessel D, Gamulin M, Kulis T, Kaneva R, Usmani N, Singhal S, Slavov C, Mitev V, Parliament M, Claessens F, Joniau S, Van den Broeck T, Larkin S, Townsend PA, Aukim-Hastie C, Gago-Dominguez M, Castelao JE, Martinez ME, Roobol MJ, Jenster G, van Schaik RHN, Menegaux F, Truong T, Koudou YA, Xu J, Khaw KT, Cannon-Albright L, Pandha H, Michael A, Thibodeau SN, McDonnell SK, Schaid DJ, Lindstrom S, Turman C, Ma J, Hunter DJ, Riboli E, Siddiq A, Canzian F, Kolonel LN, Le Marchand L, Hoover RN, Machiela MJ, Cui Z, Kraft P, Amos CI, Conti DV, Easton DF, Wiklund F, Chanock SJ, Henderson BE, Kote-Jarai Z, Haiman CA, Eeles RA; Profile Study; Australian Prostate Cancer BioResource (APCB); IMPACT Study; Canary PASS Investigators; Breast and Prostate Cancer Cohort Consortium (BPC3); PRACTICAL (Prostate Cancer Association Group to Investigate Cancer-Associated Alterations in the Genome) Consortium; Cancer of the Prostate in Sweden (CAPS); Prostate Cancer Genome-wide Association Study of Uncommon Susceptibility Loci (PEGASUS); Genetic Associations and Mechanisms in Oncology (GAME-ON)/Elucidating Loci Involved in Prostate Cancer Susceptibility (ELLIPSE) Consortium. Association analyses of more than 140,000 men identify 63 new prostate cancer susceptibility loci. Nat Genet. 2018 Jul;50(7):928-936. doi: 10.1038/s41588-018-0142-8. Epub 2018 Jun 11. PMID 29892016
- [Background] Zheng SL, Sun J, Wiklund F, Smith S, Stattin P, Li G, Adami HO, Hsu FC, Zhu Y, Balter K, Kader AK, Turner AR, Liu W, Bleecker ER, Meyers DA, Duggan D, Carpten JD, Chang BL, Isaacs WB, Xu J, Gronberg H. Cumulative association of five genetic variants with prostate cancer. N Engl J Med. 2008 Feb 28;358(9):910-9. doi: 10.1056/NEJMoa075819. Epub 2008 Jan 16. PMID 18199855
- [Background] Shi Z, Platz EA, Wei J, Na R, Fantus RJ, Wang CH, Eggener SE, Hulick PJ, Duggan D, Zheng SL, Cooney KA, Isaacs WB, Helfand BT, Xu J. Performance of Three Inherited Risk Measures for Predicting Prostate Cancer Incidence and Mortality: A Population-based Prospective Analysis. Eur Urol. 2021 Mar;79(3):419-426. doi: 10.1016/j.eururo.2020.11.014. Epub 2020 Nov 28. PMID 33257031
- [Background] Wu Y, Yu H, Li S, Wiley K, Zheng SL, LaDuca H, Gielzak M, Na R, Sarver BAJ, Helfand BT, Walsh PC, Lotan TL, Cooney KA, Black MH, Xu J, Isaacs WB. Rare Germline Pathogenic Mutations of DNA Repair Genes Are Most Strongly Associated with Grade Group 5 Prostate Cancer. Eur Urol Oncol. 2020 Apr;3(2):224-230. doi: 10.1016/j.euo.2019.12.003. Epub 2020 Jan 14. PMID 31948886
- [Background] Wu Y, Yu H, Zheng SL, Na R, Mamawala M, Landis T, Wiley K, Petkewicz J, Shah S, Shi Z, Novakovic K, McGuire M, Brendler CB, Ding Q, Helfand BT, Carter HB, Cooney KA, Isaacs WB, Xu J. A comprehensive evaluation of CHEK2 germline mutations in men with prostate cancer. Prostate. 2018 Jun;78(8):607-615. doi: 10.1002/pros.23505. Epub 2018 Mar 9. PMID 29520813

DOCUMENTS (3):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT05295407/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT05295407/SAP_001.pdf
  • Informed Consent Form (2021-11-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT05295407/ICF_002.pdf